CLINICAL TRIAL: NCT01339260
Title: A Phase III Multicenter, Randomized, Double-blind, Double-dummy, Active-controlled, Parallel Group Study of the Efficacy and Safety of Oral Netupitant Administered in Combination With Palonosetron and Dexamethasone Compared to Oral Palonosetron and Dexamethasone for the Prevention of Nausea and Vomiting in Cancer Patients Receiving Moderately Emetogenic Chemotherapy
Brief Title: An Efficacy and Safety Study of Oral Netupitant and Palonosetron for the Prevention of Nausea and Vomiting
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Helsinn Healthcare SA (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NETU-08-18
Record Dates: First submitted 2011-04-19; First posted 2011-04-20 (Estimated); Results first posted 2014-11-26 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2014-11

CONDITIONS: Chemotherapy-Induced Nausea and Vomiting
MeSH Terms: conditions — Vomiting | interventions — netupitant, palosentron drug combination; Palonosetron; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Netupitant and Palonosetron+dexamethasone-cycle 1 (Experimental): Oral netupitant/palonosetron (300 mg/0.50 mg) hard capsule with oral dexamethasone (12 mg), both given on Day 1, prior to each scheduled chemotherapy cycle
  Interventions: Drug: Netupitant and Palonosetron; Drug: Dexamethasone
- Palonosetron+dexamethasone-cycle 1 (Active Comparator): Oral palonosetron 0.50 mg (Aloxi) with oral dexamethasone (20 mg) both given on Day 1, prior to each scheduled chemotherapy cycle
  Interventions: Drug: Palonosetron; Drug: Dexamethasone
- Netupitant and Palonosetron+dexamethasone-multicycle extension (Experimental): Oral netupitant/palonosetron (300 mg/0.50 mg) hard capsule with oral dexamethasone (12 mg), both given on Day 1, prior to each scheduled chemotherapy cycle
  Interventions: Drug: Netupitant and Palonosetron; Drug: Dexamethasone
- Palonosetron+dexamethasone-multicycle extension (Active Comparator): Oral palonosetron 0.50 mg (Aloxi) with oral dexamethasone (20 mg) both given on Day 1, prior to each scheduled chemotherapy cycle
  Interventions: Drug: Palonosetron; Drug: Dexamethasone

INTERVENTIONS:
Drug: Netupitant and Palonosetron
  Arms: Netupitant and Palonosetron+dexamethasone-cycle 1; Netupitant and Palonosetron+dexamethasone-multicycle extension
Drug: Palonosetron
  Arms: Palonosetron+dexamethasone-cycle 1; Palonosetron+dexamethasone-multicycle extension
Drug: Dexamethasone

SUMMARY:
NETU-08-18 is a two-arm clinical study assessing efficacy and safety of a single oral dose of netupitant and palonosetron, two antiemetic drugs, versus oral palonosetron, both given with oral dexamethasone. The objective of the study is to demonstrate that netupitant and palonosetron are more effective than palonosetron alone, to prevent nausea and vomiting induced by moderately emetogenic cancer chemotherapy after administration of repeated cycles of chemotherapy.

DETAILED DESCRIPTION:
NETU-08-18 is a two-arm clinical study assessing efficacy and safety of a single oral dose of netupitant and palonosetron, two antiemetic drugs, versus oral palonosetron, both given with oral dexamethasone. Study is organised in two phases: cycle-1 and a multi-cycle extension. Safety assessment is performed separately in cycle 1 (arm 1 and arm 2) and in multi-cycle extension (arm 3 and arm 4).

ELIGIBILITY:
Inclusion Criteria:

* Naïve to cytotoxic chemotherapy. Previous biological or hormonal therapy will be permitted.
* Scheduled to receive first course of an anthracycline and cyclophosphamide containing moderately emetogenic chemotherapy (MEC) regimen for the treatment of a solid malignant tumor: cyclophosphamide I.V. (500 to 1500 mg/m2) and I.V. doxorubicin (more or equal to 40 mg/m2) or cyclophosphamide I.V. (500 to 1500 mg/m2) and I.V. epirubicin (more or equal to 60 mg/m2).
* If scheduled to receive chemotherapy agents of minimal to low emetogenic potential they could be given on any day.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2.
* Female patients of either non-childbearing potential or child-bearing potential with a commitment to use contraceptive methods throughout the clinical trial
* Hematologic and metabolic status adequate for receiving a moderately emetogenic regimen based on laboratory criteria (Total Neutrophils,Platelets, Bilirubin, Liver enzymes, Serum Creatinine or Creatinine Clearance)

The following inclusion criteria must be checked prior inclusion at each cycle of the Multiple-Cycle Extension:

* Participation in the study during the next cycle of chemotherapy is considered appropriate by the investigator Satisfactory study compliance in the preceding cycle of chemotherapy and related study procedures.
* Scheduled to receive the same chemotherapy regimen as cycle 1
* Adequate hematologic and metabolic status as defined for cycle 1

Exclusion Criteria:

* If female, pregnant or lactating.
* Current use of illicit drugs or current evidence of alcohol abuse.
* Scheduled to receive any highly emetogenic chemotherapy (HEC) from Day 1 to Day 5 or moderately emetogenic chemotherapy (MEC) from Day 2 to Day 5 following the allowed MEC regimen.
* Received or is scheduled to receive radiation therapy to the abdomen or the pelvis within 1 week prior to Day 1 or between Days 1 to 5 in cycle 1.
* Any vomiting, retching, or mild nausea within 24 hours prior to Day 1.
* Symptomatic primary or metastatic central nervous system (CNS) malignancy.
* Active peptic ulcer disease, gastrointestinal obstruction, increased intracranial pressure, hypercalcemia, an active infection or any uncontrolled medical condition (other than malignancy) that, in the opinion of the investigator, may confound the results of the study, represent another potential etiology for emesis and nausea (other than chemotherapy-induced nausea and vomiting, CINV) or pose unwarranted risks in administering the study drugs to the patient.
* Known hypersensitivity or contraindication to 5-HT3 receptor antagonists or dexamethasone.
* Previously received a neurokin-1 (NK1) receptor antagonist
* Participation in a clinical trial involving oral netupitant administered in combination with palonosetron.
* Any investigational drugs taken within 4 weeks prior to Day 1 of cycle 1, and/or is scheduled to receive any investigational drug during the study.
* Systemic corticosteroid therapy at any dose within 72 hours prior to Day 1 of cycle 1.
* Scheduled to receive bone marrow transplantation and/or stem cell rescue therapy.
* Any medication with known or potential antiemetic activity within 24 hours prior to Day 1 of cycle 1
* Scheduled to receive any strong or moderate inhibitor of cytocrome P450 3A4 (CYP3A4) or its intake within 1 week prior to Day 1.
* Scheduled to receive any of the following CYP3A4 substrates: terfenadine, cisapride, astemizole, pimozide.
* Scheduled to receive any CYP3A4 inducer or its intake within 4 weeks prior to Day 1.
* History or predisposition to cardiac conduction abnormalities, except for incomplete right bundle branch block.
* History of risk factors for Torsade de Point (heart failure, hypokalemia, family history of Long QT Syndrome).
* Severe cardiovascular diseases, including myocardial infarction within 3 months prior to Day 1, unstable angina pectoris, significant valvular or pericardial disease, history of ventricular tachycardia, symptomatic Congestive Heart Failure (CHF) New York Heart Association (NYHA) class III-IV, and severe uncontrolled arterial hypertension.
* Any illness or condition that, in the opinion of the investigator, may confound the results of the study or pose unwarranted risks in administering the investigational product to the patient.
* Concurrent medical condition that would preclude administration of dexamethasone such as systemic fungal infection or uncontrolled diabetes.

The following exclusion criteria must be checked prior inclusion at each cycle of the Multiple-Cycle Extension:

* If female, pregnant or lactating
* Active infection or uncontrolled disease except for malignancy.
* Started any of the restricted medications.
* Any vomiting, retching, or mild nausea within 24 hours prior to Day 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1455 (Actual)
Dates: Start 2011-04; Primary Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (172):
- United States (28):
  - Anniston Oncology/Regional Medical Center, Anniston, Alabama
  - Northwest Alabama Cancer Center, Muscle Shoals, Alabama
  - Genesis Cancer Centre, Hot Springs, Arkansas
  - Compassionate Cancer Care Medical Group Inc, Corona, California
  - Compassionate Cancer Centre Medical Group, Fountain Valley, California
  - American Institute of Research, Los Angeles, California
  - Facey Medical Group, Mission Hills, California
  - Compassionate Cancer Care Medical Group, Riverside, California
  - American Institute of Research, Whittier, California
  - Denver Health and Hospital Authority, Denver, Colorado
  - Palm Beach Institute of Hematology and Oncology, Boynton Beach, Florida
  - Baptist Cancer Institute, Jacksonville, Florida
  - Deaconess Clinic Downtown, Evansville, Indiana
  - Floyd Memorial Cancer Center of Indiana, New Albany, Indiana
  - Kentucky Cancer Clinic, Hazard, Kentucky
  - The John R Marsh Cancer Center, Hagerstown, Maryland
  - Fallon Clinic at Worcester Medical Center, Worcester, Massachusetts
  - Duke University Medical Center, Durham, North Carolina
  - Piedmont Hematology Oncology Associates PA, Winston-Salem, North Carolina
  - Tri-County Hematology and Oncolgy Associates Inc., Massillon, Ohio
  - Signal Point Clinical Research Center LLC, Middletown, Ohio
  - Charleston Cancer Center, Charleston, South Carolina
  - Charleston Hematology Oncology, Charleston, South Carolina
  - Wellmont Medical Associates-Oncology and Hematology, Bristol, Tennessee
  - Cancer Specialists of South Texas, P.A., Corpus Christi, Texas
  - The University of Texas Health Center, Tyler, Texas
  - Northern Utah Associates Hematology / Oncology, Ogden, Utah
  - Northwest Medical Specialties, Tacoma, Washington
- Argentina (9):
  - Hospital Italiano de Cordoba, Córdoba
  - Clínica Universitaria Reina Fabiola (Universidad Católica de Córdoba), Córdoba
  - Instituto Oncológico de Córdoba - Sanatorio Aconcagua, Córdoba
  - Centro Oncológico Integral (COI), Mar del Plata
  - Centro Oncologico de Integracion Regional (COIR), Mendoza
  - Instituto Médico CER [Oncology], Quilmes
  - Sanatorio Parque, Rosario
  - Centro Medico San Roque, San Miguel de Tucumán
  - ISIS Clinica Especializada, Santa Fe
- Belarus (6):
  - Bobruisk Interregional Oncological Dispensary, Babruysk
  - Brest Regional Oncological Dispensary, Brest
  - Gomel Regional Clinical Oncological Dispensary, Brest
  - Minsk city Clinical Oncological Dispensary [Oncology], Minsk
  - State institution N.N. Alexandrov Republican Scientific and Practical Center of Oncology and Medical Radiology, Minsk
  - Mogilev Regional Oncological Dispensary [Oncology], Mogilev
- Brazil (12):
  - OXION-Medicina Oncológica, Belo Horizonte
  - Centro de Pesquisas Clínicas em Oncologia, Cachoeiro de Itapemirim
  - IPCEM - Centro de Ciências da Saúde - Universidade de Caxias, Caxias do Sul
  - Hospital Araújo Jorge, Goiânia
  - Clinica de Neoplasias do Litoral, ItajaÃ
  - Clinica De Oncologia De Porto Alegre S S Ltda, Porto Alegre
  - Hospital Moinhos de Vento, Porto Alegre
  - Instituto Ribeirãopretano de Combate ao Cancer, Ribeirão Preto
  - Oncotrat Oncologia Medica Ltda [Oncology], Rio de Janeiro
  - Nucleo de Oncologia da Bahia, Salvador Bahia
  - Hospital Santa Cruz, São Paulo
  - Casa de Saude Santa Marcelina, São Paulo
- Bulgaria (12):
  - SHATO "Sveti Mina", Blagoevgrad
  - MHAT Dr. Tota Venkova [Oncology], Gabrovo
  - Specialized Hospital for Active Treatment of Oncology, Haskovo
  - UMHAT ""Dr. Georgi Stranski"" Dept. Medical Oncology, Pleven
  - UMHAT "Sveti Georgi" [Clinic of Oncology and Hematology], Plovdiv
  - District Dispensery with Stationary - Sofia District, Sofia
  - UMHAT "Tsaritsa Yoanna - ISUL" Ltd.Medical Oncology Clinic, Sofia
  - Specialized Hospital for Active Treatment in Oncology, Sofia
  - Specialized Hospital for Active Treatment of Onclogy Diseases - Sofia City, Sofia
  - Complex Oncology Centre, Stara Zagora
  - COC - Veliko Tarnovo Dept. Medical Oncology, Veliko Tarnovo
  - Comprehensive Cancer Center - Vratsa Dept. of Palliative Care, Vratsa
- Croatia (9):
  - Županijska bolnica Cakovec, Čakovec
  - Klinicki bolnicki centar Osijek [Oncology], Osijek
  - Opca bolnica Pula [Odjel za onklologiju], Pula
  - KBC Rijeka [Gastroenterology], Rijeka
  - Opca bolnica Varazdin [Odjel za hem.onko i klin.imun.], Varaždin
  - Opca Bolnica Zadal Ulica, Zadar
  - Klinički bolnički centar Zagreb [Oncology], Zagreb
  - Klinicka bolnica [Sestre milosrdnice], Zagreb
  - Klinika za tumore [Odjel za kemoter. i internisticku onkolog, Zagreb
- Germany (11):
  - Klinik und Poliklinik für Onkologie und Hämatologie Universitatsmedizin Charite Mitte, Berlin
  - Gynäkologische Arztpraxis, Berlin
  - OncoResearch Lerchenfeld UG, Hamburg
  - Schwerpktprxs gynäkolog Onkologie Prof. Dr. Diel, Dr. Gebert, Mannheim
  - Rotkreuzklinikum [München], München
  - Tumorzentrum Munchen Sued - Städtisches Klinikum [Hämato-, Onkologie + Palliativmed], München
  - Staedtisches Krankenhaus Muenchen Neuperlach, München
  - OncoPRO GbR Dr. R. Dengler, Dr. A. Kröber Gesellschaft für klinische Studien in der ambulanten Hämatologie und Onkologie, Regensburg
  - Universitätsklinikum Tübingen, Tübingen
  - Praxis Dr. G. Dresemann, Velen
  - Onkologische Gemeinschaftspraxis Dr. med M. Perker / PF Dr. med M. Sandherr, Weilheim
- Hungary (8):
  - Semmelweis Egyetem Kútvölgyi Klinikai Tömb, Budapest
  - Fővárosi Önkormányzat Uzsoki utcai Kórház, Budapest
  - Petz Aladár Megyei Oktató Kórház [Onkoradiológiai Oszt, Győr
  - Bács-Kiskun Megyei Önkormányzat Kórháza, Szegedi, Kecskemét
  - Borsod-Abaúj-Zemplén Megyei Kórház és Egyetemi Oktató Kórház, Miskolc
  - Josa Andras Oktato Korhaz [Onkologiai Osztaly], Nyíregyháza
  - Pécsi Tudományegyetem Klinikai Köpont, Pécs
  - Jasz-Nagykun-Szolnok Megyei Hetenyi Geza Korhaz, Szolnok
- India (13):
  - HCG - Multy Speciality Hospital, Ahmedabad
  - Hemato-Oncology Clinic Ahmedabad Pvt Ltd, Ahmedabad
  - Sujan Surgical Cancer Hospital and Amracvati Cancer Foundation, Amravati
  - Sri Venkateshwara Hospital [Medical Oncology], Bangalore
  - Apollo Speciality Hospital, Chennai
  - Dr. Kamahshi Memorial Hospital [Oncology], Chennai
  - BIBI General Hospital & Cancer Centre [Oncology], Hyderabad
  - Yashoda B-Block Hospital, Hyderabad
  - B.P.Poddar Hospital and Medical Research Ltd, Kolkata
  - Apollo Gleneagles Hospitals Kolkata, Kolkata
  - Shatabdhi Superspeciality Hospital, Nashik
  - Grant Medical Foundation - Ruby Hall Clinic, Pune
  - City Cancer Centre [Surgical and Medical Oncology], Vijayawada
- Italy (5):
  - Fondazione Poliambulanza Istituto Ospedaliero, Brescia
  - Ospedale Vito Fazzi, ASL Lecce, Lecce
  - Presidio Ospedaliero "Alessandro Manzoni", AO Provincia di Lecco, Lecco
  - Ospedale Sacro Cuore e Don Calabria - Negrar, Negrar
  - Ospedale S.Carlo di Potenza [U.O. di Oncologia Medica], Potenza
- Mexico (5):
  - Centro Oncologico De Chihuahua, Chihuahua City
  - Hospital de Jesus, México
  - Centro Medico Quirurgico, México
  - OCA Hospital/Monterrey International Research Center, Monterrey
  - Centro Regiomontano de Investigación Clínica, Monterrey
- Poland (10):
  - Bialostockie Centrum Onkologii im. M.Sklodowskiej-Curie, Bialystok
  - Wojewodzki Szpital Zespolony w Elblagu, Oddzial Onkologiczny, Elblag
  - Niepubliczny Specjalist. Onkol. Zaklad Opieki Zdrowotnej, Kościerzyna
  - Wojewodzki Szpital Specjalistyczny im. M.Kopernika, Lodz
  - Olsztynski Osrodek Onkologiczny "KOPERNIK", Olsztyn
  - Szpital Rejonowy im. dr J. Rostka w Raciborzu, Racibórz
  - Wojewodzki Szpital Specjalistyczny im. J. Korczaka, Słupsk
  - Centrum Onkologii - Instytut im. Marii Sklodowskiej - Curie, Warsaw
  - NZOZ Magodent - Centrum Medczyne Ostrobramska, Warsaw
  - Szpital Wojewodzki w Lomzy im. Kardynala S. Wyszynskiego, Łomża
- Romania (10):
  - Spitalul Judetean de Urgenta "Dr. Constantin Opris" Baia-Mare [Oncologie Medicala], Baia Mare
  - Spitalul Universitar de Urgenta Elias [Oncologie Medicala], Bucharest
  - Spitalul Clinic CF nr.2 Bucuresti [Oncologie Medicala], Bucharest
  - Spitalul Universitar de Urgenta Bucuresti, Bucharest
  - Institutul Oncologic "Prof. Dr. Alex. Trestioreanu" [Sectia Clinica Radioterapie II], Bucharest
  - Oncolab - Oncology Center Craiova, Craiova
  - Institutul Regional de Oncologia, Iași
  - Spitalul Municipal Onesti [Sectia Oncologie Medicala], Onești
  - Spitalul Clinic Judetean Mures, Tg Mures
  - Oncomed SRL, Timișoara
- Russia (22):
  - GUZ Arkhangelsk Regional Clinical Oncological Dispensary, Arkhangelsk
  - Ivanovo Regional Oncological Dispensary [Chemotherapy], Ivanovo
  - GAUZ Republic Clinical Oncology Dispensary of Ministry of Health of Republic Tatarstan, Kazan'
  - GOU VPO Krasnoyarsk State Medical University n.a. prof. V.F., Krasnoyarsk
  - GUZ Lipetsk Regional Oncology Dispensary [General Oncology], Lipetsk
  - GUZ Regional Oncology Dispensary #2, Magnitogorsk
  - Russian Cancer Research Center, Moscow
  - SBHI of Moscow City Oncology Clinical Hospital #62, Moscow
  - MBUZ City Clinical Hospital #1, Novosibirsk
  - FGBU Medical Radiology Scientific Center, Obninsk
  - GUZ Perm Regional Oncology Dispensary, Perm
  - GUZ Pyatigorsk Oncology Dispensary [Outpatient Department], Pyatigorsk
  - GOU VPO - Ryazan State Med. Univer. n.a. I.I.Pavlov based Ryazan Regio, Ryazan
  - GUZ "Leningrad Regional Oncology Dispensary", Saint Petersburg
  - City Oncology Dispensary, Saint Petersburg
  - GOU VPO Saint-Petersburg State Medical University n.a. acad., Saint Petersburg
  - St. Petersburg Clinical Oncology Dispesary - 3rd Gynecology D, Saint Petersburg
  - FGU Research Institute of Oncology n.a. N.N.Petrov of Rosmed, Saint Petersburg
  - GUZ Samara Regional Clinical Oncology Dispensary, Samara
  - Stavropol Regional Clinical Oncology Dispensary, Stavropol
  - GBUZ - Clinical Oncology Dispensary of MoH of Republic Bahkortostan, Ufa
  - GUZ Republican Clinical Oncological Dispensary of public, Ufa
- Ukraine (12):
  - Komunalnyi "Cherkaskyi oblasnyi onkolohichnyi dyspanser" Cherkaskoi oblasnoi rady, oblasnyi onkokhimioterapevtychnyi tsentr, m. Cherkasy, Cherkasy
  - Komunalnyi likuvalno-profilaktychnyi zaklad "Chernigivskyi, Chernihiv
  - Chmelnytskyi Regional Clinical Oncology Centre [Oncology], Chmelnytskyi
  - Komunalnyizaklad Miska bahatoprofilna klinichna likarnia #4, Dnipropetrovks
  - Donetskyi oblasnyi protypukhlynnyi tsentr, Donetsk
  - Kharkivskyi oblasnyi onkologichnyi klinichnyi tsentr, Kharkiv
  - Kyirskyi Miskyi klinichnyi onkolohichnyi tsentr, Kyiv
  - KZ KOR Kyivskyi oblasnyi onkologichnyi dyspanser, Kyiv
  - Lvivskyi derzhavnyi onkologichnyi regionalnyi likuvalno diahnostychyi tsentr, Lviv
  - Odeska oblasna klinichna likarnia, Odesa
  - Poltavskyi oblasnyi klinichnyi onkolohichnyi dyspanser Pol, Poltava
  - Zakarpatskyi oblasnyi klinichnyi onkodyspanser, Uzhhorod

REFERENCES:
- [Derived] Schwartzberg L, Karthaus M, Rossi G, Rizzi G, Borroni ME, Rugo HS, Jordan K, Hansen V. Fixed combination of oral NEPA (netupitant-palonosetron) for the prevention of acute and delayed chemotherapy-induced nausea and vomiting in patients receiving multiple cycles of chemotherapy: Efficacy data from 2 randomized, double-blind phase III studies. Cancer Med. 2019 May;8(5):2064-2073. doi: 10.1002/cam4.2091. Epub 2019 Apr 9. PMID 30968588
- [Derived] Rugo HS, Rossi G, Rizzi G, Aapro M. Efficacy of NEPA (netupitant/palonosetron) across multiple cycles of chemotherapy in breast cancer patients: A subanalysis from two phase III trials. Breast. 2017 Jun;33:76-82. doi: 10.1016/j.breast.2017.02.017. Epub 2017 Mar 10. PMID 28285236

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1455 patients randomized (ITT population), 1450 received study drug i.e. netupitant/palonosetron combination or palonosetron, both with dexamethasone, in cycle 1 (safety population-cycle 1), 1449 received chemotherapy and study drug (FAS), 1286 received study drug in multi-cycle extension (safety population-multi-cycle extension)
Groups:
- Netupitant and Palonosetron Plus Dexamethasone: Oral netupitant/palonosetron (300 mg/0.50 mg) hard capsule with oral dexamethasone, both given on Day 1, prior to each scheduled chemotherapy cycle
  Netupitant and Palonosetron
  Dexamethasone
- Palonosetron Plus Dexamethasone: Oral palonosetron 0.50 mg (Aloxi) with oral dexamethasone both given on Day 1, prior to each scheduled chemotherapy cycle
  Palonosetron
  Dexamethasone
Period: Cycle 1
Arm/Group | Netupitant and Palonosetron Plus Dexamethasone | Palonosetron Plus Dexamethasone
Started | 726 (Intent-To-Treat: randomized patients) | 729 (Intent-To-Treat: randomized patients)
Safety Population | 725 (Patients receiving netupitant/palonosetron combination) | 725 (Patients receiving palonosetron)
Full Analysis Set | 724 (Patients receiving chemotherapy and randomized to netupitant/palonosetron combination) | 725 (Patients receiving chemotherapy and randomized to palonosetron)
Completed | 719 | 719
Not Completed | 7 | 10
Period: Multi-cycle Extension
Arm/Group | Netupitant and Palonosetron Plus Dexamethasone | Palonosetron Plus Dexamethasone
Started | 635 (Patients scheduled to netupitant/palonosetron combination) | 651 (Patients scheduled to palonosetron)
Safety Population | 635 (Patients receiving netupitant/palonosetron combination) | 651 (Patients receiving palonosetron)
Completed | 449 (Patients completing at least number of cycles they were scheduled to) | 458 (Patients completing at least number of cycles they were scheduled to)
Not Completed | 186 | 193

BASELINE CHARACTERISTICS:
Population: Safety population ie patients receiving either netupitant/palonosetron combination or palonosetron, both plus dexamethasone
Groups:
- Total: Total of all reporting groups
Arm/Group | Netupitant and Palonosetron Plus Dexamethasone | Palonosetron Plus Dexamethasone | Total
Number analyzed (Participants) | 725 | 725 | 1450
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (10.66) | 54.1 (10.65) | 53.9 (10.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 711 | 711 | 1422
  Male | 14 | 14 | 28
Race/Ethnicity, Customized [Number; unit: participants]
  White | 574 | 579 | 1153
  Black | 1 | 3 | 4
  Asian | 101 | 103 | 204
  Hispanic | 46 | 36 | 82
  Other | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Complete Response (CR) Defined as no Emesis, no Rescue Medication, at Cycle 1
Time Frame: 25-120 hours
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | Netupitant and Palonosetron Plus Dexamethasone | Palonosetron Plus Dexamethasone
Number analyzed (Participants) | 724 | 725
percentage of responders | 76.9 [73.7 to 79.9] | 69.5 [66.1 to 72.8]
Statistical Analysis 1: Comparison: Netupitant and Palonosetron Plus Dexamethasone vs Palonosetron Plus Dexamethasone; The null hypothesis was rejected if the 2 sided p value from the Cochran Mantel Haenszel test was less than or equal to 0.050 and in the right direction i.e., the Odds Ratio (OR) was in favor of netupitant/palonosetron. Power was 90%; Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel — If superiority of netupitant/palonosetron was established for the CR delayed, CR acute and then CR overall at cycle 1 were to be tested according to a hierarchical procedure;no adjustment for multiplicity was needed.The a priori threshold was 0.050; Odds Ratio (OR) = 1.48, 95% CI 2-sided [1.16 to 1.87] — Cochran Mantel Haenszel (CMH) test including treatment, age class and region as strata. All missing data were to be imputed as treatment failures

2. Secondary Outcome: Percentage of Patients With Complete Response (CR) Defined as no Emesis, no Rescue Medication at Cycle 1
Time Frame: 0-24 hours
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | Netupitant and Palonosetron Plus Dexamethasone | Palonosetron Plus Dexamethasone
Number analyzed (Participants) | 724 | 725
percentage of responders | 88.4 [85.9 to 90.5] | 85.0 [82.2 to 87.4]
Statistical Analysis 1: Comparison: Netupitant and Palonosetron Plus Dexamethasone vs Palonosetron Plus Dexamethasone; CR in the acute phase was to be tested using the same 2 sided CMH test as for the primary endpoint. netupitant/palonosetron combination was to be considered superior to palonosetron in the acute phase if the 2 sided p value from the CMH was less than or equal to 0.050 and in the right direction; Test type: Superiority or Other; p = 0.047, Cochran-Mantel-Haenszel — If the null hypothesis for CR delayed was rejected, analysis of the first key secondary endpoint CR acute was to be performed. Since the analysis was performed according to a hierarchical procedure, no further adjustment for multiplicity was needed; Cochran Mantel Haenszel (CMH) test including treatment, age class and region as strata. All missing data were to be imputed as treatment failures; Odds Ratio (OR) = 1.37, 95% CI 2-sided [1.0 to 1.87]

3. Secondary Outcome: Percentage of Patients With Complete Response (CR) Defined as no Emesis, no Rescue Medication, at Cycle 1
Time Frame: 0-120 hours
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | Netupitant and Palonosetron Plus Dexamethasone | Palonosetron Plus Dexamethasone
Number analyzed (Participants) | 724 | 725
percentage of responders | 74.3 [71.0 to 77.4] | 66.6 [63.1 to 70.0]
Statistical Analysis 1: Comparison: Netupitant and Palonosetron Plus Dexamethasone vs Palonosetron Plus Dexamethasone; CR in the overall phase was to be tested using the same 2 sided CMH test as for the primary endpoint. netupitant/palonosetron combination was to be considered superior to palonosetron in the overall phase if the 2 sided p value from the CMH was less than or equal to 0.050 and in the right direction; Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel — If the null hypothesis for CR acute was rejected, analysis of the 2nd key secondary endpoint CR overall was to be performed. Since the analysis was performed according to a hierarchical procedure, no further adjustment for multiplicity was needed; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.47, 95% CI 2-sided [1.17 to 1.85]

ADVERSE EVENTS:
Time Frame: Period from time of informed consent signature until 21 days post study drugs (Day 1 of the last cycle). Upon Investigator's judgment, all non resolved, non serious Adverse Events (AEs) beyond this date could have been followed for an additional 14 days
Description: AEs are presented separately for cycle 1 and for multi-cycle extension (i.e. without Cycle 1), consistent with Analysis Plan and Clinical Study Report
Arm/Group | Netupitant and Palonosetron+Dexamethasone-cycle 1 | Palonosetron+Dexamethasone-cycle 1 | Netupitant and Palonosetron+Dexamethasone-multicycle Extension | Palonosetron+Dexamethasone-multicycle Extension
Serious Adverse Events (participants affected / at risk) | 13/725 | 12/725 | 23/635 | 15/651
Other Adverse Events (participants affected / at risk) | 551/725 | 507/725 | 533/635 | 527/651
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Netupitant and Palonosetron+Dexamethasone-cycle 1 (N=725) | Palonosetron+Dexamethasone-cycle 1 (N=725) | Netupitant and Palonosetron+Dexamethasone-multicycle Extension (N=635) | Palonosetron+Dexamethasone-multicycle Extension (N=651)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 3 | 6 | 4
Leukopenia (Blood and lymphatic system disorders) | 2 | 0 | 1 | 2
Neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 6 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 1
Cytotoxic cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0 | 1 | 0
Central venous catheterisation (Surgical and medical procedures) | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 1
General physical health deterioration (General disorders) | 0 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0
Device relatet infections (Infections and infestations) | 0 | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fibrin D dimer increased (Investigations) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Arterial thrombosis limb (Vascular disorders) | 0 | 0 | 1 | 0
Venous recanalisation (Vascular disorders) | 0 | 0 | 0 | 1
Venous thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
Cardiac failure acute (Cardiac disorders) | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Catheterisation venous (Surgical and medical procedures) | 0 | 1 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 1 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 2 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Netupitant and Palonosetron+Dexamethasone-cycle 1 (N=725) | Palonosetron+Dexamethasone-cycle 1 (N=725) | Netupitant and Palonosetron+Dexamethasone-multicycle Extension (N=635) | Palonosetron+Dexamethasone-multicycle Extension (N=651)
Leukopenia (Blood and lymphatic system disorders) | 96 | 90 | 138 | 141
Neutropenia (Blood and lymphatic system disorders) | 173 | 182 | 226 | 238
Asthenia (General disorders) | 59 | 50 | 70 | 69
Fatigue (General disorders) | 47 | 38 | 49 | 49
Headache (Nervous system disorders) | 64 | 52 | 53 | 57
Alopecia (Skin and subcutaneous tissue disorders) | 253 | 253 | 152 | 151
Anaemia (Blood and lymphatic system disorders) | 26 | 24 | 47 | 41
Constipation (Gastrointestinal disorders) | 31 | 26 | 27 | 33
Diarrhoea (Gastrointestinal disorders) | 13 | 10 | 33 | 21
Nausea (Gastrointestinal disorders) | 22 | 27 | 27 | 35
Decreased appetite (Metabolism and nutrition disorders) | 25 | 32 | 28 | 42
Hyperglycaemia (Metabolism and nutrition disorders) | 24 | 25 | 45 | 43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor and investigator(s) agree that no publications discussing trials' results will occur until release of final report. Sponsor has no objections if the investigators publish study results, however the investigator is requested to contact the sponsor before publishing, to prevent premature disclosure of data and is not intended as a restrictive measure concerning results or opinions of investigators.